CLINICAL TRIAL: NCT04291612
Title: SEntinel Lymph Node Endometrial Cancer Trial: A Prospective Multicenter International Single-Arm Observational Trial (SELECT)
Brief Title: Observational Study of Women With Endometrial Cancer Who Receive the Standard Treatment for Their Disease
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-067
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer; Endometrioid Adenocarcinoma; Endometrial Cancer Stage I
Keywords: Endometrial Cancer; Endometrioid Adenocarcinoma; 20-067; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma, Endometrioid | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1: Participants will have endometrioid adenocarcinoma histological diagnosis with planned surgical treatment including hysterectomy in combination with SLN biopsy.
- Part 2: Participants will have undergone surgery and bilateral sentinel lymph node mapping (negative for malignancy)
  Interventions: Other: Physical exam

INTERVENTIONS:
Other: Physical exam — Part 2 participants will be prospectively followed clinically for relapse for 30 months from the date of surgery for physical examination at post-ops visits.
  Groups: Part 2

SUMMARY:
This study is being done to find out how often endometrial cancer recurs after the standard treatment as well as how often the standard treatment results in a lymphedema.

ELIGIBILITY:
Screening Inclusion Criteria:

* ECOG performance status 0-1 or KPS ≥ 70%
* Age ≥ 18 years
* Endometrioid adenocarcinoma histologic diagnosis on endometrial biopsy or dilatation and curettage
* No evidence of extrauterine disease, or suspicious pelvic lymph nodes, or distant metastases, or cervical invasion on pre-operative conventional imaging studies (Pelvic +/- Abdomen CT or MRI or sonogram, or body PET scan) and physical examination (uterine confined by exam and imaging )
* Suitable candidate for surgery
* Planned surgical treatment including hysterectomy in combination with SLN biopsy and a bilateral salpingo-oophorectomy
* No history of second primary cancer (invasive or in situ) within the past 5 years, not including non-melanoma skin cancer
* Approved and signed informed consent
* No history of neoadjuvant chemotherapy or radiotherapy for endometrial cancer
* No history of prior pelvic or abdominal radiotherapy

Screening Exclusion Criteria:

* Extrauterine disease, or gross lymph node involvement, or cervical invasion suspected on pre-operative imaging studies and physical examination (disease not uterine confined clinical stage > I)
* Contraindication for SLN mapping
* The planned treatment is not surgery, or the surgical treatment does not include hysterectomy in combination with SLN biopsy and a bilateral salpingo-oophorectomy

Eligibility Inclusion Criteria

Patients will be classified in the study cohort (part 2; n=182) according to surgical treatment received, final post hysterectomy and staging pathologic report, and planned adjuvant treatment. The inclusion criteria are specified below.

Study Cohort (n=182)

A patient will be enrolled in the study cohort if all the following criteria are met:

* At surgery, the patient must undergo:

  * Hysterectomy
  * Bilateral salpingo-oophorectomy, unless already performed (including allowing unilateral salpingo-oophorectomy if unilateral salpingo-oophorectomy already performed)
  * Bilateral pelvic SLN mapping (bilateral sentinel nodes are negative for malignancy)
* On the final pathologic report, the patient must have a diagnosis of:

  * Stage I intermediate-risk endometrial endometrioid cancer (Grade 1 or Grade 2 with ≥ 50% myometrial invasion or Grade 3 with <50% myometrial invasion, including non-invasive disease)
  * Negative pelvic peritoneal cytology
* Adjuvant treatment as recommended by the multidisciplinary team must be as follows:

  * No adjuvant treatment, or
  * Intravaginal radiation only

Eligibility Exclusion Criteria

* There is intra-operative detection of extra-uterine disease or grossly involved lymph nodes
* Presence of any positive pelvic nodes including micrometastasis and isolated tumor cells (ITC)
* Hysterectomy is not performed
* Bilateral salpingo-oophorectomy is not performed, unless already performed (unilateral salpingo-oophorectomy is allowed if unilateral salpingo-oophorectomy already performed)
* Failed unilateral or bilateral SLN mapping
* Patient undergoes a complete unilateral or bilateral pelvic lymphadenectomy
* Patient undergoes a radical type C hysterectomy
* Stage IA endometrioid cancer Grade1 or 2 and myometrial invasion <50%
* Stage IB Grade 3 endometrioid cancer
* Non-endometrioid histology: Serous, clear cell, carcinosarcoma, undifferentiated, or de-differentiated histology noted on final hysterectomy pathology
* Empty unilateral or bilateral sentinel lymph nodal packet(s)
* Positive peritoneal cytology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or a member of the research teams. If the investigator is a member of the treatment team, s/he will screen their patients' medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study. The principal investigators may also screen the medical records of patients with whom they do not have a treatment relationship for the limited purpose of identifying patients who would be eligible to enroll in the study, and to record appropriate contact information in order to approach these patients regarding the possibility of enrolling in the study. Patients identified in this manner would subsequently be approached for study enrollment after consultation with their treating physician.
Sampling Method: Probability Sample
Enrollment: 1715 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of pelvic/non-vaginal recurrence at 36 months | 36 months
  Participants will be assessed every 6 (+/- 2) months for 36 months through routine physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Abu-Rustum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (19):
- United States (13):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - University of Miami (Data Collection Only), Miami, Florida
  - Miami Cancer Institute Baptist Health South Florida, Miami, Florida
  - ADVENTHEALTH (Data collection only), Orlando, Florida
  - Mayo Clinic (Data Collection and Data Analysis), Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
- Charles University and General University Hospital (Data Collection Only), Prague, Czechia
- Italy (4):
  - OSPEDALE MICHELE E PIETRO (Data Collection Only), Ferrera
  - UNIVERSITY OF MILANO-BICOCCA, ITALY (Data Collection), Milan
  - FONDAZIONE POLICLINICOUNIVERSITARIO A. GEMELLI, ITALY (Data Collection Only), Roma
  - L'Azienda Sanitaria Universitaria Friuli Centrale, Udine
- OSLO UNIVERSITY HOSPITAL,RIKSHOPITALET (Data Collection Only), Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Grassi T, Mariani A, Cibula D, Soliman PT, Suman VJ, Weaver AL, Pedra Nobre S, Weigelt B, Glaser GE, Cappuccio S, Abu-Rustum NR. A prospective multicenter international single-arm observational study on the oncological safety of the sentinel lymph node algorithm in stage I intermediate-risk endometrial cancer (SELECT, SEntinel Lymph node Endometrial Cancer Trial). Int J Gynecol Cancer. 2020 Oct;30(10):1627-1632. doi: 10.1136/ijgc-2020-001698. Epub 2020 Jul 22. PMID 32699021
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org